CLINICAL TRIAL: NCT07273058
Title: Effect of High-Intensity Interval Training Intervention on Post-Stroke Fatigue in Chronic Stroke Survivors: A Pilot Randomized Clinical Trial
Brief Title: Effect of HIIT on Post-Stroke Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr HUANG Mei Zhen, Assistant professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20241002001
Record Dates: First submitted 2025-09-16; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT (Experimental)
  Interventions: Behavioral: HIIT
- MICT (Active Comparator)
  Interventions: Behavioral: MICT
- Stretching (Active Comparator)
  Interventions: Behavioral: stretching

INTERVENTIONS:
Behavioral: HIIT — The HIIT intervention will consist of a 3-minute warm-up, a 25-minute main exercise, and a 2-minute cool-down. The main exercise will include four 4-minute high-intensity intervals, each interspersed with a 3-minute low-intensity recovery period. Participants will attend three supervised sessions per week over a 12-week period.
  Arms: HIIT
Behavioral: MICT — The MICT intervention will include a 3-minute warm-up, 25 minutes of continuous exercise performed at a moderate intensity, and a 2-minute cool-down. Participants will attend three supervised sessions per week over a 12-week period.
  Arms: MICT
Behavioral: stretching — The stretching intervention will consist of 30 minutes of whole-body stretching. Participants will attend three sessions per week over a 12-week period.
  Arms: Stretching

SUMMARY:
This study aims to investigate the effect of high-intensity interval training (HIIT) on fatigue severity among individuals with chronic stroke. Participants will be randomly assigned to the HIIT group, the moderate-intensity continuous training (MICT) group, or the stretching group (active control). Each group will participate in supervised exercise sessions three times per week over a 12-week period, totaling 36 sessions. Outcome assessments will be conducted at baseline, mid-intervention (week 6), post-intervention (week 12), and follow-up (week 20). The primary outcome will be fatigue severity. Secondary outcomes will include inflammatory biomarkers and additional health-related indicators.

ELIGIBILITY:
Inclusion criteria:

* Age of 40-80 years;
* a history of ischemic stroke resulting in unilateral limb impairment 6-60 months prior to consent to participate in the pilot trial;
* a stable medical condition;
* a subjective feeling of fatigue, defined as a period of apparent fatigue, decreased energy, increased need for rest, or fatigue out of proportion to physical activity for at least 2 weeks during the past month;
* ability to communicate with the investigators and lack of significant cognitive deficits;
* able to walk for 10 meters with or without a walking aid.

Exclusion criteria:

* An FSS score of < 4 (20);
* other neurological conditions;
* other musculoskeletal comorbidities that would prevent safe participation in exercises;
* a medical diagnosis of significant cardiovascular, pulmonary, or metabolic disease(s);
* signs or symptoms indicative of significant cardiovascular, pulmonary, or metabolic disease(s) during the previous 3 months;
* severe lower limb spasticity (Ashworth Scale score ≥ 3);
* Botulinum toxin use in the affected lower limb within the past six months;
* current or previous use of drugs intended to resolve post-stroke fatigue;
* active engagement in other stroke rehabilitation trials.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Eligibility rate (%) | Through study completion, an average of 12 weeks.
Recruitment rate (number of participants per month) | Through study completion, an average of 12 weeks.
Compliance with HIIT (%) | From baseline to week 12
Fidelity to the HIIT protocol (%) | From baseline to week 12
Retention of the intervention (%) | From baseline to week 12
Adverse events (number of events) | From baseline to week 12
Acceptability (qualitative) | At week 12

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | Blinded assessors will conduct evaluations at baseline, week 12 , and week 20.
  The FSS consists of 9 items rated on a 7-point Likert scale from 1 (highly disagree) to 7 (highly agree). Higher scores indicate greater fatigue severity.
Multidimensional Fatigue Inventory (MDI) | Blinded assessors will conduct evaluations at baseline, week 12 , and week 20.
  The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report questionnaire designed to assess fatigue across five dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation, and Reduced Activity. Each subscale contains 4 items rated on a 5-point Likert scale. Higher scores indicate greater fatigue. The total score ranges from 20 to 100.
Short Form-36 Health Survey (SF-36) | Blinded assessors will conduct evaluations at baseline, week 6, and week 12.
  The SF-36 includes 36 items and one additional item assessing perceived change in health over time. Each domain is scored on a scale from 0 to 100, with higher scores indicating better health status.
Inflammatory biomarkers | Blinded assessors will conduct evaluations at baseline, week 6, and week 12.
  Inflammatory biomarkers will be quantified using enzyme-linked immunosorbent assay (ELISA) kits obtained from commercial suppliers, following the manufacturer's instructions.

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Blinded assessors will conduct evaluations at baseline, week 12 , and week 20.
  The HADS consists of 14 items, divided into two subscales: anxiety (HADS-A) and depression (HADS-D), each containing 7 items. Each item is scored on a 4-point Likert scale (0-3), resulting in subscale scores ranging from 0 to 21. Higher scores indicate greater severity of anxiety or depression.
Pittsburgh Sleep Quality Index (PSQI) | Blinded assessors will conduct evaluations at baseline, week 12 , and week 20.
  The PSQI is consists of 19 items grouped into seven components. Each component is scored from 0 to 3, yielding a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Stroke Self-Efficacy Questionnaire (SSEQ) | Blinded assessors will conduct evaluations at baseline, week 12 , and week 20.
  The SSEQ is a 13-item self-report scale assessing stroke survivors' confidence in performing daily activities and managing post-stroke challenges. Each item is rated from 0 (not at all confident) to 4 (very confident). Total score ranges from 0 to 52. Higher scores indicate greater self-efficacy.
Fugl-Meyer Motor Assessment-Lower Extremity | Blinded assessors will conduct evaluations at baseline, week 12 , and week 20.
  To assess motor recovery, Fugl-Meyer Motor Assessment-Lower Extremity will be used, it score rangefrom 0 to 34; a high score is indicative of good motor recovery
6-Minute Walk Test | Blinded assessors will conduct evaluations at baseline, week 12 , and week 20.
  Walking endurance will be assessed using the 6-Minute Walk Test. The participants will be allowed to use assistive devices, which will be documented and kept consistent across all of the time points.
Physical Activity Enjoyment Scale (PAES) | Blinded assessors will conduct evaluations at week 6 and at week 12.
  The PAES will be used to measure the participants' exercise enjoyment (score range: 0-56). A high score indicates a high level of activity enjoyment.
Behavioral Regulation In Exercise Questionnaire (BREQ-2) | Blinded assessors will conduct evaluations at week 1, week 12, and week 20.
  The BREQ-2 includes 19 items. Each item is rated on a 5-point Likert scale ranging from 0 ("not true for me") to 4 ("very true for me"). Higher scores reflect higher exercise motivation.
Mini Balance Evaluation Systems Test (MiniBEST) | Blinded assessors will conduct evaluations at baseline, week 12 , and week 20.
  The Mini-BESTest consists of 14 items, including the Timed Up and Go test, with a maximum total score of 28 points. Higher scores indicate better balance performance.
Short Physical Performance Battery (SPPB) | Blinded assessors will conduct evaluations at baseline, week 12 , and week 20.
  The SPPB comprises three components: balance tests (including side-by-side, semi-tandem, and tandem stances), a gait speed test, and a five-times sit-to-stand test. Each component is scored on a scale from 0 to 4, with a total possible score ranging from 0 to 12. Higher scores indicate better physical performance.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided